CLINICAL TRIAL: NCT04068233
Title: Impact of Pacing Mode and Diastolic Function on Cardiac Output
Acronym: PADIAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kepler University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Clemens Steinwender, Head of the Department of Cardiology, Kepler University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 01/2019
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Diastolic Function; Cardiac Output; Pacemaker Stimulation Mode; Stroke Volume; AV Block
Keywords: Diastolic function; Cardiac output; Pacemaker stimulation mode; Stroke volume
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Intervention Model Description: Each patient will represent their own control, as both pacing modes (asynchronous and synchronous) are applied in each patient.
Who Masked: Participant, Investigator
Masking Description: It is decided by coin tossing which pacing mode is programmed first (randomization). Sonographer and patient are both blinded to the pacing mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eligible patients - pacing mode sequence 1 (Experimental): Echo assessment of parameters of diastolic function, systolic function, and atrial function. Then, the stroke volume and cardiac output are measured during AV-asynchronous and AV-synchronous pacemaker stimulation: AV-synchronous pacing mode first, then AV-dyssynchronous pacing mode.
  Interventions: Other: Pacemaker stimulation mode
- Eligible patients - pacing mode sequence 2 (Experimental): Echo assessment of parameters of diastolic function, systolic function, and atrial function. Then, the stroke volume and cardiac output are measured during AV-asynchronous and AV-synchronous pacemaker stimulation: AV-dyssynchronous pacing mode first, then AV-synchronous pacing mode.
  Interventions: Other: Pacemaker stimulation mode

INTERVENTIONS:
Other: Pacemaker stimulation mode — Echocardiographic indices are measured during AV asynchronous and AV synchronous pacemaker stimulation.

SUMMARY:
Background It is known from previous research that in patients with complete AV (atrioventricular) block and pacemaker stimulation stroke volume and cardiac output are higher with AV-synchronous than with AV-dyssynchronous pacing. However, the extent to which patients profited from AV-synchronous stimulation varied substantially.

Aim of the study Aim of this study is to systematically analyze the impact of diastolic function and other echo parameters on the difference of stroke volumes/cardiac output between AV-synchronous and AV-dyssynchronous pacing modes.

Methods Patients fulfilling the entry criteria will be enrolled (two-chamber pacemaker of any vendor eligible) in this monocentric, prospective, interventional study. Baseline data will be collected with a standardized questionnaire. During an echo examination, parameters of diastolic, systolic and atrial function will be assessed. Then, the stroke volume/cardiac output will be measured twice in each patient, once with AV-synchronous and once with AV-dyssynchronous pacing. Therefore, each patient will represent their own control. It will be randomized (coin tossing) which stimulation mode is first and which is second (sonographer and patient will be blinded). Descriptive statistics will be applied and regression models will be fitted to explore the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able and willing to give informed consent and is above the age of 18.
* Patient is implanted with a dual chamber pacemaker system for at least 6 weeks.
* Patient is in sinus rhythm on the day of recruitment.
* Patient has a ventricular pacing rate exceeding 90%.
* Upon initial device interrogation, parameters are within normal ranges.
* Calculated battery life is more than 1 year.

Exclusion Criteria:

* Patient is not in sinus rhythm on the day of echo examination.
* Intrinsic ventricular activation on the day of echo examination.
* Relevant shunt on the atrial, ventricular or pulmonary level.
* Moderate or severe heart valve dysfunction (stenosis or regurgitation).
* Presence of other medical devices that may interact with the pacemaker system.
* Women who are pregnant or breast feeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Effect of left ventricular diastolic function on the change of cardiac output between AV-synchronous and AV-asynchronous pacing modes. | During echo examination.
  Echo parameters of diastolic function.

SECONDARY OUTCOMES:
Effect of left ventricular systolic function on the change of cardiac output between AV-synchronous and AV-asynchronous pacing modes. | During echo examination.
  Echo parameters of systolic function.
Effect of atrial function on the change of cardiac output between AV-synchronous and AV-asynchronous pacing modes. | During echo examination.
  Echo parameters of atrial function.
Effect of baseline characteristics on the change of cardiac output between AV-synchronous and AV-asynchronous pacing modes. | During echo examination.
  Demographic variables and co-morbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Steinwender, Assoc. Prof., MD, Principal Investigator — Kepler University Hospital, Department of Cardiology
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blessberger H, Kammler J, Kellermair J, Kiblboeck D, Nahler A, Hrncic D, Saleh K, Schwarz S, Reiter C, Fellner A, Eppacher C, Sheldon TJ, Steinwender C. Impact of pacing mode and different echocardiographic parameters on cardiac output (PADIAC). Front Cardiovasc Med. 2023 May 17;10:1185518. doi: 10.3389/fcvm.2023.1185518. eCollection 2023. PMID 37265566